CLINICAL TRIAL: NCT07172542
Title: High Risk of Death or Disability in Brain Hemorrhage: Role of Spot Sign and Secondary Markers
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier de Gonesse (Other)
Responsible Party: Sponsor
Other Study IDs: 0125_REANIMATION_SPOT-TARGET
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Intracerebral Hemorrhage; Cerebral Hemorrhage; Stroke; Brain Injuries
MeSH Terms: conditions — Cerebral Hemorrhage; Stroke; Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (4):
- Intracerebral Hemorrhage Without Spot Sign or Secondary Morphological Marker
- Spot Sign Only
- Spot Sign With a Secondary Morphological Marker
- Single Secondary Morphological Marker Without Spot Sign

SUMMARY:
This study looks at patients with brain hemorrhage to see if a special sign on brain scans, called the "Spot Sign," combined with other scan features, can predict a higher risk of death or disability. By comparing patient outcomes with existing prediction scores, the study aims to understand whether these scan markers provide extra value in identifying patients at higher risk.

ELIGIBILITY:
Inclusion Criteria:

* Spontaneous intracerebral hemorrhage confirmed by contrast-enhanced CT scan.
* Follow-up CT scan performed within 24 to 48 hours.

Non-inclusion Criteria :

* Absence of initial contrast-enhanced CT or follow-up CT.
* Hematoma due to trauma, epidural hematoma (EDH), subdural hematoma (SDH), or subarachnoid hemorrhage (SAH).

Exclusion Criteria:

* Patient deceased before the initial contrast-enhanced CT.
* Major missing clinical data.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Source Population: Patients hospitalized for hemorrhagic stroke (spontaneous ICH) in the neurology department, with an available initial contrast-enhanced CT scan.
  Target Population: Patients with non-traumatic spontaneous intracerebral hemorrhage (ICH).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Hematoma Expansion within 48 Hours: Increase of more than 6 mL or over 30% between the initial CT and the follow-up CT (PREDICT study criterion) and/or Occurrence of Death Within the First Month | 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de Gonesse, Gonesse, France, France